CLINICAL TRIAL: NCT03175185
Title: Psychiatric Assessment Of Parents Of Children With Attention Deficit Hyperactivity Disorder
Brief Title: Psychiatric Assessment Of Parents Of Children With ADHD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Osman Mohammed Elnady Ellisy, Dr, Assiut University
Other Study IDs: 17100221
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents of children with ADHD: 100 parents of 50 children who were diagnosed with ADHD and
- Parent of children without ADHD: 100 parents of 50 children who are ADHD free as a control group

SUMMARY:
The aim of this study is to carry out a psychological evaluation for the parents of children diagnosed with attention deficit hyperactivity disorder (ADHD) and parents of children without ADHD as control to detect any psychological problems in those of children with ADHD . These problems may be a precipitating factor to cause ADHD in their child or have a genetic predisposition to be passed to their children. On the other hand these psychological problems may be caused by the difficulties they encounter in raising their ADHD child. The exact relation needs more researches and to be more investigated.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children diagnosed with ADHD according to the American Psychiatric Association's Diagnostic and Statistical Manual (DSM-V).
* Children are between 4 and 16 years of age for both sexes.
* Children with normal IQ > 70%.
* Parents are able to give informed consent and able to complete the research assessments.

Exclusion Criteria:

* Parents having chronic debilitating diseases e.g. chronic liver cirrhosis.
* Parents were participating in other clinical research.
* Refusal to participate.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The people participating in this study will be 100 parents of 50 children who were diagnosed with ADHD and 100 parents of 50 children who are ADHD free as a control group recruited from outpatient clinic of Assiut University hospital.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Psychiatric Assessment of the parents | 2 years
  Detection of personality disorders, anxiety and depressive symptoms

IPD SHARING:
Plan to Share IPD: Undecided